CLINICAL TRIAL: NCT04446897
Title: Treatment of Chronic Medium-severe Periodontitis With Mesenchymal Stem Cells Predifferentiated in Osteogenic Direction Immobilised on a Biodegradable Carrier
Brief Title: Treatment of Chronic Medium-severe Periodontitis With Mesenchymal Stem Cells Predifferentiated in Osteogenic Direction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC(periodontitis)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Periodontitis, Chronic
Keywords: Periodontitis; Mesenchymal stem cells
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cells (Experimental): standard treatment according to clinical protocols plus mesenchymal stem cells
  Interventions: Biological: mesenchymal stem cells; Other: standard treatment
- standard treatment (Active Comparator): standard treatment according to clinical protocols
  Interventions: Other: standard treatment

INTERVENTIONS:
Biological: mesenchymal stem cells — autologous mesenchymal stem cells
  Arms: mesenchymal stem cells
Other: standard treatment — standard treatment according to clinical protocols

SUMMARY:
Treatment of chronic medium-severe periodontitis with mesenchymal stem cells and mesenchymal stem cells predifferentiated in osteogenic direction

DETAILED DESCRIPTION:
The bone defect will be filled with a porous membrane based on bone collagen measuring 5x5 mm or more with mesenchymal stem cells and mesenchymal stem cells predifferentiated in osteogenic direction

ELIGIBILITY:
Inclusion Criteria:

- chronic medium-severe periodontitis

Exclusion Criteria:

* pregnancy
* breast-feeding
* acute and chronic infectious diseases: HIV, viral hepatitis, tuberculosis
* mental disorders

Ages: 70 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
number of patients cured | 1 month
  number of patients cured

CONTACTS AND LOCATIONS:
Overall Officials: Igor Volotovski, Prof, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering; Sergey Rubnikovich, Prof, Study Director — Head of the Department of Prosthodontics of BMAPE
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus